CLINICAL TRIAL: NCT05784974
Title: An Open-label, Single-center, Phase II Study of Cadonilimab Monotherapy as Neoadjuvant Therapy for Resectable II-IIIA Squamous Cell Lung Cancer
Brief Title: Cadonilimab Monotherapy as Neoadjuvant Therapy for Resectable II-IIIA Squamous Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23K004-001
Record Dates: First submitted 2023-03-10; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (Experimental): Participants receive two cycles of Cadonilimab as neoadjuvant therapy prior to surgery; followed by surgery; followed by standard adjuvant chemotherapy +/- adjuvant Cadonilimab for 6 months.
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — 15 mg/kg via intravenous infusion on Day 1 of each 21-day cycle.

SUMMARY:
Cadonilimab, a tetravalent bispecific antibody targeting PD-1 and CTLA-4, is designed to retain the efficacy benefit of combination of PD-1 and CTLA-4 and improve on the safety profile of the combination therapy. The aim of this study is to evaluate the efficacy and safety of Cadonilimab monotherapy as neoadjuvant therapy for patients with resectable stage II-IIIA squamous cell lung cancer.

ELIGIBILITY:
Key Inclusion Criteria:

Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 2. Have previously untreated and pathologically confirmed resectable Stage II-IIIA Squamous cell lung cancer.

Have at least one measurable lesion per RECIST 1.1 assessed by investigator. Have adequate organ function.

Key Exclusion Criteria:

Mixed adenocarcinoma and small cell lung cancer histology. Patients with other active malignancies within 5 years prior to enrollment. Known active autoimmune diseases. Use of immunosuppressive agents within 14 days prior to the first dose of study treatment.

Presence of other uncontrolled serious medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) Rate | After surgery (approximately 7 weeks)
  defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate | After surgery (approximately 7 weeks)
  defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy
Complete (R0) Resection Rate | After surgery (approximately 7 weeks)
  defined as the percentage of participants achieving complete surgical resection following completion of neoadjuvant therapy.
Objective Response Rate (ORR) | At the end of 2 cycles of neoadjuvant therapy (each cycle is 21 days)
  defined as the percentage of participants having complete response or partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Disease Free Survival (DFS) | Up to approximately 5 years
  defined as the time from the first dose of study drug to disease progression per RECIST 1.1 that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first.
Adverse Events (AEs) | From the first dose of neoadjuvant treatment until 90 days after the last dose of adjuvant treatment

IPD SHARING:
Plan to Share IPD: No